CLINICAL TRIAL: NCT02522806
Title: Endometrial Local Injury Before First IVF : Evaluation of Pregnancy Rate
Acronym: BEONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1408062; 2014-A01003-44 (Other: ANSM)
Record Dates: First submitted 2015-08-12; First posted 2015-08-13 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Sterility, Female
Keywords: Endometrial biopsy; previous ovarian hyperstimulation cycle; first IVF; antagonist protocol; clinical pregnancy rate
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Endometrial biopsy (EB) between J17 and J22 of previous ovarian hyperstimulation cycle.
  Interventions: Procedure: endometrial biopsy
- Group B (No Intervention): none endometrial biopsy

INTERVENTIONS:
Procedure: endometrial biopsy — Endometrial biopsy (EB) between J17 and J22 of previous ovarian hyperstimulation cycle
  Arms: Group A

SUMMARY:
In spite of all progress realized in the field of assisted reproduction the pregnancy rate by In vitro fertilization (IVF) in France, across indications, is only 23% after IVF cycle.

Different causes may account for these failures and that, during all stages of pregnancy.

Recent studies have investigated an essential step in fecundation : uterine receptivity. Some teams have shown that a lot of immunological factors would have very significant in this step, by them possible expression in this process. Other studies looked at genes modulation, essential to implantation, with endometrium manipulation, simple, such as endometrial biopsy (EB). The last findings published on this subject, but after 2 IVF failures, are most encouraging because the pregnancy rate for these teams after just endometrial local injury (EB after 2 IVF failures) is well above their usual pregnancy rate. Some teams have focused on immunoassay of endometrial biopsy, in order to profile uterine receptivity and suggest with results, suitable treatment for each patient (ongoing study).

EB is quick, easy, make in a simple consultation and with a low cost, contrary to immunological study, which depend of ultra-specialized laboratories and therefore with an important cost.

ELIGIBILITY:
Inclusion Criteria:

* Only first IVF
* Acceptance of protocol by patient after free and complete information and signature of consent.
* Anti-Mullerian Hormone (AMH ) greater than 1
* Member or eligible to social security system
* Availabilities for a follow up 2 or 12 months.

Exclusion Criteria:

* Known intolerance of proposed treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2014-09-23 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
number of Early pregnancy | Day 28
  Early pregnancy is defined by beta human chorionic gonadotropin (HCG)>100 mIU/ml defined by at least one rate of beta HCG>100 on the 3 possible dosages after embryo transfer (if first dosage negative or >100 : stop, if first dosage positive but <100 : Second dosing, if >100 or less than first result : stop, otherwise third dosing).
  Endometrial biopsy (diameter : 1mm ; length : 5mm) with use a pipelle, in the second part of the cycle between J17 and J22 during cycle before IVF

SECONDARY OUTCOMES:
Number of middle pregnancy | 5 weeks of amenorrheas.
  Middle pregnancy is defined by an intra uterine gestation sac on echography of 5 or 6 weeks of amenorrheas.
Number of late pregnancy | 12 weeks of amenorrheas.
  Late pregnancy is defined by an intra uterine evolutionary pregnancy on echography of 12 weeks of amenorrheas.
number of Live birth | delivery
number of patient with endometrial chronic infection | Day 22 of previous cycle of IVF
  Presence of endometrial chronic infection is measured by histopathologic analysis of biopsy
number of patient with pain | Day 22 of previous cycle of IVF
  Pain is estimated by visual analogue scale note at the end of biopsy (day 22 of previous cycle of IVF)
number of patient with endometrial acute infection | Day 24 of previous cycle of IVF
  An endometrial acute infection is defined by pelvic spontaneous pain and/or leucorrhoea, abnormal metrorrhagia and/or fever appearing after biopsy.
number of patient with uterine perforation | Day 22 of previous cycle of IVF
  An uterine perforation is defined by intense pain at the time of the biopsy or in the days to come and/or leucorrhoea, abnormal metrorrhagia and/or fever.

CONTACTS AND LOCATIONS:
Overall Officials: Anne GENOD, MD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No